CLINICAL TRIAL: NCT00470262
Title: Effects of PPAR Ligands on Ectopic Fat Accumulation and Inflammation in Subjects With Impaired Glucose Tolerance
Brief Title: Effects of PPAR Ligands on Ectopic Fat Accumulation and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ENDA-020-06S; 09-0710 (Other: COMIRB)
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Metabolic Syndrome X; Prediabetic State
Keywords: fatty acid oxidation complex; fenofibrate; Inflammation; Peroxisome Proliferator-Activated Receptors; pioglitazone; Prediabetic State; insulin resistance
MeSH Terms: conditions — Metabolic Syndrome; Prediabetic State; Inflammation; Insulin Resistance | interventions — Fenofibrate; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fenofibrate 145 mg PO QD and Pioglitazone 45 mg PO QD (Other): Treatment with pioglitazone and fenofibrate in subjects with pre diabetes
  Interventions: Drug: Fenofibrate 145mg PO QD; Drug: Pioglitazone 45 mg PO QD
- Fenofibrate 145 mg PO QD (Other): Treatment with fenofibrate in subjects with pre diabetes
  Interventions: Drug: Fenofibrate 145mg PO QD

INTERVENTIONS:
Drug: Fenofibrate 145mg PO QD — Subjects will be randomized to either fenofibrates or combination of both fenofibrate and pioglitazone
  Other Names: Tricor
Drug: Pioglitazone 45 mg PO QD — Subjects will be randomized to either fenofibrate 145 mg PO QD or a combination of both fenofibrate 145 mg PO QD and pioglitazone 45 mg PO QD
  Other Names: Actos
  Arms: Fenofibrate 145 mg PO QD and Pioglitazone 45 mg PO QD

SUMMARY:
The relationship between obesity and insulin resistance is known, however the mechanism(s) associating obesity with insulin resistance is not well understood. Inflammation and accumulation of fat in non fat tissue (like muscle) are conditions found on obesity which could be the potential link between obesity and insulin resistance. This study is designed to test the effects of two different drugs on numerous features of the obesity and insulin resistance in subjects with impaired glucose tolerance. Impaired glucose tolerance is a condition where blood sugar is too high after drinking a sugary drink containing 75 grams of sugar. Impaired glucose tolerant subjects are insulin resistant and at risk of developing diabetes. The drugs to be used are fenofibrate and pioglitazone. Fenofibrate is used to reduce the amount of fat (triglycerides) in the blood while pioglitazone is routinely used to make the body more sensitive to insulin in patients with diabetes. The purpose of this study is to compare the effects of either of these two medications (pioglitazone and fenofibrate) alone or the combination of both on fat accumulation in body (muscle) and inflammation. The amount of fat accumulation in muscle is thought to affect insulin sensitivity. In addition, the changes in the level of proteins produced by fat tissues will be studied in response to the two medications in this study. These proteins are thought to be involved in diabetes and insulin resistance.

These studies are designed to examine fundamental clinical mechanisms underlying the metabolic syndrome and diabetes.

DETAILED DESCRIPTION:
The correlation between obesity, inflammation and ectopic fat accumulation is well recognized; however, the mechanism(s) responsible for obesity induced insulin resistance is not well understood. The investigators will focus on lipotoxicity and inflammation as the link between obesity and insulin resistance. The factors leading to inflammation and ectopic lipid accumulation in obesity and the best intervention to reverse this pathophysiology are not clear. In this study, the investigators will examine inflammation in adipose tissue and muscle lipid mechanism in response to Peroxisome Proliferator Activated Receptors (PPAR) and ligands have synergistic anti-inflammatory effects in adipose tissue and activation of PPAR and decrease muscle lipid oxidation and redistribution of lipid from muscle to adipocytes respectively. The combination of both medications will be particularly effective in reducing inflammation and muscle lipid accumulation.

In this study, IGT subjects will be randomized to treatment with PPAR ligand (fenofibrate), PPAR ligand (pioglitazone) or combination of both for 10 weeks. Baseline studies will include assessment of body composition, insulin sensitivity, muscle and fat biopsies. All studies will be repeated after treatment with fenofibrate, pioglitazone or combination of both.

Specific Aims (SA) are as follows:

SA 1. Insulin sensitivity and Intramyocellular lipid (IMCL) from muscle biopsy specimens will be measured in response to different treatments (PPAR , and combination of both ligands).

SA 2. The rate of fatty acid oxidation and the number of mitochondria in muscle will be measured in response to PPAR ligands.

SA 3. The anti-inflammatory effects of PPAR and ligands will be studied by the measurement of the number of adipose tissue macrophages and the rate of macrophages apoptosis in fat biopsy specimens. In addition, the plasma levels and expression of proinflammatory proteins will be studied in response to different treatment.

SA 4. The rate of SUMOylation of PPAR (a novel mechanism regulating anti-inflammatory effects of PPAR ligands) will be studied in response to PPAR , ligand or combination of both.

These studies are designed to examine fundamental clinical mechanisms underlying the metabolic syndrome and diabetes.

Potential Impact on Veterans Health Care: The national obesity/diabetes epidemic is magnified in the VA, and the cost of caring for these patients is enormous. This study will provide data on the mechanism of action of these drugs, which will improve the investigators' understanding of these drugs, impaired glucose tolerance, and treatment of metabolic syndrome. From the clinical perspective, this study uses drugs to treat patients with IGT, which is rapidly becoming recognized as a "disease" because of its association with coronary artery disease risk factors, and because of its high rate of progression to T2DM. If these drugs were shown to improve the care of patients, then they would eventually be a cost savings to the VA, either by choosing the less expensive drug, or by using the drug that delays the progression of the disease, and improves the care of the patient by preventing complications.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance and/or impaired fasting glucose and/or metabolic syndrome
* Age 18-65
* BMI 28-38

Exclusion Criteria:

* Renal insufficiency: creatinine.1.4
* Liver disease: ALT.2x normal, congestive heart failure, history of documented coronary artery disease, concomitant use HMG CoA-reductase inhibitors (statins)
* Concurrent use of ASA, steroids and other anti-inflammatory agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-01; Primary Completion 2012-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neda Rasouli, MD, Principal Investigator — VA Eastern Colorado Health Care System, Denver
Locations (1):
- VA Eastern Colorado Health Care System, Denver, Denver, Colorado, United States

REFERENCES:
- [Derived] Ipsen EO, Madsen KS, Chi Y, Pedersen-Bjergaard U, Richter B, Metzendorf MI, Hemmingsen B. Pioglitazone for prevention or delay of type 2 diabetes mellitus and its associated complications in people at risk for the development of type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 19;11(11):CD013516. doi: 10.1002/14651858.CD013516.pub2. PMID 33210751

RESULTS

PARTICIPANT FLOW:
Groups:
- Fenofibrate: Treatment with fenofibrate 145mg PO QD
- Piolitazone 45 mg PO QD + Fenofibrate 145mg PO QD: Pioglitazone and Fenofibrate: Subjects will be randomized to a combination of both fenofibrate(145mg PO QD) and pioglitazone 45 mg PO QD
Period: Overall Study
Arm/Group | Fenofibrate | Piolitazone 45 mg PO QD + Fenofibrate 145mg PO QD
Started | 15 | 12
Completed | 13 | 12
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fenofibrate 145 mg PO QD: Treatment fenofibrate 145 mg PO QD in subjects with pre diabetes
- Fenofibrate 145 mg PO QD and Pioglitazone 45mg PO QD: Treatment with Fenofibrate 145 mg PO QD and Pioglitazone 45mg PO QD in subjects with pre diabetes
- Total: Total of all reporting groups
Arm/Group | Fenofibrate 145 mg PO QD | Fenofibrate 145 mg PO QD and Pioglitazone 45mg PO QD | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.69 (8.46) | 44.67 (11.49) | 46.76 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 9 | 2 | 11
Region of Enrollment [Number; unit: participants]
  United States | 15 | 12 | 27
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.06 (3.51) | 33.93 (3.49) | 33.99 (3.43)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Insulin sensitivity was measure through frequently sampled intravenous glucose tolerance test. Subjects presented to research center fasting. Blood samples were collected at -21, -11, and -1 minutes. At time t=0 initiates the start of the IVGTT and the injection of glucose into the non-sampling arm. The glucose dose was calculated as 11.4g/m2 of body surface area, given as a 50% dextrose solution. This glucose injection was administered over 60 seconds or less. At time t=20 minutes, an insulin dose of 0.04u/kg was administered over 30 seconds. Blood samples were collected at times t=2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 19, 22, 23, 24, 25, 27, 30, 40, 50, 70, 90, 100, 120, 140, 160, and 180. If blood sugar did not return to a steady state the test was continued to t= 210 or t= 240.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg*kg^-1*min^-1
Groups:
- Fenofibrate 145mg PO QD: Treatment with fenofibrate in subjects with pre diabetes
- Fenofibrate 145 mg PO QD + Pioglitazone: Treatment with fenofibrate and pioglitazone in subjects with pre diabetes
Arm/Group | Fenofibrate 145mg PO QD | Fenofibrate 145 mg PO QD + Pioglitazone
Number analyzed (Participants) | 13 | 12
mg*kg^-1*min^-1
  pre | 1.48 (0.64) | 1.73 (0.75)
  post | 1.89 (0.88) | 2.93 (1.3)

2. Secondary Outcome: IMCL
Description: Intramyocellular lipid was measured using immunohistochemistry (using oil Red O staining) in muscle biopsy specimens. Oil red O-stained muscle sections were magnified with an Olympus Provis (Tokyo, Japan) light microscope, and images were digitally captured by using a connected charge-coupled device camera (Sony, Tokyo, Japan). Fiber-typed and oil red O-stained fibers were matched. The oil red O staining intensity of either type 1 or 2 muscle fibers was quantified using National Institutes of Health Image program (http://rsb.info.nih.gov/nih-image/). By adjusting a density threshold, the software was set to recognize the presence of one fat droplet only if its highlighted surface was exceeding 0.40 μm2 or larger. Muscle lipid content was calculated by total area of lipid droplets in a given muscle fiber divided by the total area of the same fiber. The mean number of fibers analyzed per sample was 40 for type 1 and 2 muscle fibers
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: % of lipid area stained
Groups:
- Fenofibrate 145mg PO QD + Pioglitazone 45mg PO BID: Treatment with pioglitazone and fenofibrate in subjects with pre diabetes
Arm/Group | Fenofibrate 145mg PO QD | Fenofibrate 145mg PO QD + Pioglitazone 45mg PO BID
Number analyzed (Participants) | 13 | 12
% of lipid area stained
  pre | 3.67 (1.30) | 5.32 (0.65)
  post | 3.46 (2.36) | 2.82 (0.56)

ADVERSE EVENTS:
Groups:
- Fenofibrate 145mg PO QD: Treatment with fenofibrate 145 mg PO QD in subjects with pre diabetes
- Fenofibrate 145 mg PO QD and Pioglitazone 45 mg PO QD: Treatment with fenofibrate 145 mg PO QD and Pioglitazone 45 mg PO QD in subjects with pre diabetes
Arm/Group | Fenofibrate 145mg PO QD | Fenofibrate 145 mg PO QD and Pioglitazone 45 mg PO QD
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/12
Other Adverse Events (participants affected / at risk) | 0/15 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenofibrate 145mg PO QD (N=15) | Fenofibrate 145 mg PO QD and Pioglitazone 45 mg PO QD (N=12)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) — unrelated to study medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No